CLINICAL TRIAL: NCT00412412
Title: A Ph1 Open-Label,Dose-Escalation,Safety,PK & PD Study of CNF2024 as a Single-Agent Treatment in Subjects w/HER2- Adv Breast Cancer or in Combo w/Trastuzumab in Subjects w/HER2+ Advanced Breast Cancer
Brief Title: CNF2024 (BIIB021) HER2- (QD) HER2+ (BIW w/Herceptin) PK/PD Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Julie Morrissey, Quintiles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120BC101
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: Cancer of Breast; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients with HER2- Breast Cancer
  Interventions: Drug: CNF2024
- B (Experimental): Patients with HER2+ Breast Cancer
  Interventions: Drug: CNF2024 + trastuzumab

INTERVENTIONS:
Drug: CNF2024 — Oral doses of CNF2024 as specified in the protocol.
  Other Names: BIIB021
  Arms: A
Drug: CNF2024 + trastuzumab — Oral doses of CNF2024 as specified in the protocol Intravenous doses of trastuzumab as specified in the package insert.
  Other Names: BIIB021 (CNF2024); Herceptin (trastuzumab)
  Arms: B

SUMMARY:
The goal of this clinical research study is to study the drug CNF2024 as a single agent or in combination with trastuzumab in patients with advanced breast cancer and to:

* find the highest dose of the drug CNF2024 as a single agent or in combination with trastuzumab that can be given safely
* measure levels of CNF2024 as a single agent or in combination with trastuzumab in blood
* determine if CNF2024 as a single agent or in combination with trastuzumab can stop breast cancer cells from growing

DETAILED DESCRIPTION:
A Phase 1 Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of CNF2024 as a Single-Agent Treatment in Subjects with HER2- Advanced Breast Cancer or in Combination with Trastuzumab in Subjects with HER2+ Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria (Group A):

* Age ≥18 years at the time of informed consent.
* Male and female subjects with confirmed HER2 adenocarcinoma of the breast with advanced disease (advanced disease will be defined as metastatic disease or locally advanced disease that is surgically unresectable and considered unmanageable with standard therapies such as radiation or systemic therapies) who have had disease progression on at least one standard hormonal or chemotherapy regimen for advanced breast cancer or who have refused standard therapies.
* Evaluable disease either by measurable disease (RECIST) or nonmeasurable disease.
* ECOG ≤2.
* Required Laboratory Values:ANC ≥1500 cells/mm3,platelet count ≥100,000 cells/mm3,hemoglobin ≥9 gm/L; Glucose >3.3 mmol/L, sodium >130 mmol/L, calcium >2.0 mmol/L.
* Plasma cortisol and ACTH levels that are not suggestive of adrenal insufficiency.
* Normal electrocardiogram (ECG) with QTc ≤450 msec for men and ≤470 msec for women.
* Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to first study drug administration.

Inclusion Criteria (Group B):

* Age ≥18 years at the time of informed consent.
* Male and female subjects with confirmed HER2+ (IHC 3+ or IHC 2+/FISH+) adenocarcinoma of the breast with advanced disease that have had disease progression on at least 1 standard hormonal or chemotherapy regimen for advanced metastatic breast cancer. Advanced disease will be defined as metastatic disease or locally advanced disease that is surgically unresectable and considered unmanageable with standard therapies such as radiation or systemic therapies.
* Subjects must have progressed either within 3 months following last dose of adjuvant trastuzumab treatment or progressed following trastuzumab based therapies for metastatic disease.
* Measurable disease by RECIST or evaluable nonmeasurable disease
* ECOG ≤2.
* Required Laboratory Values: ANC ≥1500 cells/mm3,platelet count ≥100,000 cells/mm3,hemoglobin ≥9 gm/L; Glucose >3.3 mmol/L, sodium >130 mmol/L, calcium >2.0 mmol/L.
* Plasma cortisol and ACTH levels that are not suggestive of adrenal insufficiency.
* Normal ECG with QTc ≤450 msec for men and ≤470 msec for women.
* Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to first study drug administration.

Exclusion Criteria (Group A):

* Prior antitumor therapies including prior experimental agents or approved antitumor therapies, within 1 month.
* Active infection requiring intravenous (IV) antibiotic treatment.
* History of prior malignancies within the past 5 years with the exception of curatively treated basal or squamous cell carcinomas of the skin or carcinoma in situ of the cervix.
* Concurrent severe or uncontrolled diabetes and/or other medical disease
* Problems with swallowing or malabsorption.
* History of major surgery to small intestine.
* Prior treatment with Hsp90 inhibitors.
* History of central nervous system (CNS) metastasis.

Exclusion Criteria (Group B):

* Prior antitumor therapies, including prior experimental agents or approved antitumor therapies, within 1 month.
* Active infection requiring intravenous (IV) antibiotic treatment.
* History of prior malignancies within the past 5 years with the exception of curatively treated basal or squamous cell carcinomas of the skin or carcinoma in situ of the cervix.
* Concurrent severe or uncontrolled diabetes and/or other medical disease
* Problems with swallowing or malabsorption.
* History of major surgery to small intestine.
* Cardiac left ventricular function with resting ejection fraction <50%, assessed by either ECHO or MUGA.
* Prior treatment with Hsp90 inhibitors.
* Diabetes treated with insulin.
* History of CNS metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Clinical and laboratory safety assessments | 30 days after discontinuation of CNF2024 or until drug-related toxicites have returned to less than Grade 1

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Tampa, Florida
  - Research Site, New York, New York
  - Research site, Houston, Texas